CLINICAL TRIAL: NCT03360474
Title: The Implementation of a Delirium Screening and Intervention Protocol for Critically Ill Patients
Brief Title: Implementation of a Delirium Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed to a QI project
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Maria Rueda-Lara, Assistant Profesor of Clinical Psychiatry, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20170784
Record Dates: First submitted 2017-11-17; First posted 2017-12-04 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2017-11

CONDITIONS: Delirium; Cancer; Bone Marrow Ablation
MeSH Terms: conditions — Delirium; Neoplasms

STUDY DESIGN:
Intervention Model Description: Descriptive analysis will be conducted on demographic (e.g., age, gender) variables to report characteristics of the sample. The data to be collected are reflected in the attached measures. Days spent in the ICU and total days spent in the hospital will be analyzed using standard t-tests to assess difference in length of stay in ICU and overall hospitalization for 60 days prior to initiation of the delirium protocol and 60 days following the initiation of the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will be placed on the delirium screening intervention protocol arm. They will be screened for delirium twice per day. If positive, they will follow the treatment algorithm and assessed at 4 hour intervals until they reach 4 negative screens. Once 4 negative screens have been reached, they will be assessed twice daily.
  Interventions: Behavioral: Delirium Screen

INTERVENTIONS:
Behavioral: Delirium Screen — Patients who screen positive for delirium will be assessed for pain, electrolyte imbalances,infection, the use of deliriogenic medications and any issues will be resolved. Those with persistent delirium following all other intervention will be treated with antipsychotic medication.

SUMMARY:
The purpose of this project is to improve patient outcomes in individuals affected by cancer, through the implementation of a delirium screening and treatment protocol in the ICU setting. The hypothesis is that patients who receive an accurate and early diagnosis of delirium coupled with a standardized intervention protocol will demonstrate improved patient outcomes as evidenced by fewer days spent in the ICU, fewer days spent in the hospital (overall length of stay) and the need for less sedative medication throughout their ICU stay as compared to patient data prior to the implementation of a delirium protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included into the study who:

  * Are over 18 years old
  * Speak and read English
  * Are admitted to the Sylvester Comprehensive Cancer Center intensive care unit in the first 60 days following implementation of the delirium protocol; approximately 10 patients per month.
  * Patient data via electronic medical record (EMR) for all patients who were admitted to the Sylvester Comprehensive Cancer Center intensive care unit up to 60 days prior to the implementation of the delirium protocol.

Exclusion Criteria:

* This study will exclude:

  * Patients who are unable to speak and read English
  * Patients who are unable to provide written consent to participate.
  * Patient data via EMR for any patients who were admitted to the Sylvester Comprehensive Cancer Center intensive care unit prior to 60 days before to the implementation of the delirium protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
ICU Length of Stay (LOS) | 60 days
  Patient's length of stay in the ICU

SECONDARY OUTCOMES:
Overall LOS in hospital | 60 days
  Patient's length of stay in hospital
Sedation Medication | 60 days
  Total amount of sedating medication given to patient during their hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rueda-Lara, MD, Principal Investigator — SCCC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. 5th ED. Washington, DC: American Psychiatric Association; 2013.
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] McNicoll L, Pisani MA, Zhang Y, Ely EW, Siegel MD, Inouye SK. Delirium in the intensive care unit: occurrence and clinical course in older patients. J Am Geriatr Soc. 2003 May;51(5):591-8. doi: 10.1034/j.1600-0579.2003.00201.x. PMID 12752832
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] Breitbart W, Alici Y. Evidence-based treatment of delirium in patients with cancer. J Clin Oncol. 2012 Apr 10;30(11):1206-14. doi: 10.1200/JCO.2011.39.8784. Epub 2012 Mar 12. PMID 22412123
- [Background] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Background] Brummel, N., Jackson, J., Torres, R. et al: Does duration of ICU delirium predict long-term functional impairment? Am J. Respir Crit Care Med 2011; 183: A2653
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Spronk PE, Riekerk B, Hofhuis J, Rommes JH. Occurrence of delirium is severely underestimated in the ICU during daily care. Intensive Care Med. 2009 Jul;35(7):1276-80. doi: 10.1007/s00134-009-1466-8. Epub 2009 Apr 7. PMID 19350214
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Costabile S, Truman Pun B, Dittus R, Ely EW. Motoric subtypes of delirium in mechanically ventilated surgical and trauma intensive care unit patients. Intensive Care Med. 2007 Oct;33(10):1726-31. doi: 10.1007/s00134-007-0687-y. Epub 2007 Jun 5. PMID 17549455
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] 0-10 Numeric Pain Rating Scale: From McCaffery M, Pasero C. Pain: Clinical Manual, St. Louis, 1999, P. 16.
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407